CLINICAL TRIAL: NCT00416585
Title: Effects of Roaccutane on Ca, P, PTH and Vitamin D Metabolites in the Treatment
Brief Title: Effects of Roaccutane on Ca, P, PTH and Vitamin D Metabolites in the Treatment of Sever Acne
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: src-hmnm-1385
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Acne
Keywords: acne; isotretinoin; calcium. vitamin D
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

INTERVENTIONS:
Drug: isotretinoin (Roaccutane)

SUMMARY:
serum levels Ca, P, PTH and vitamin D metabolites before and after treatment with isotretinoin for sever acne

DETAILED DESCRIPTION:
few studies has been done of serum levels Ca, P, PTH and vitamin D metabolites in patients receiving isotretinoin .In this study we measured serum levels Ca, P, PTH and vitamin D metabolites before and after treatment with isotretinoin for sever acne in 30 patients . the patients had no kown skeletal, endocrine ,renal and gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* sever acne

Exclusion Criteria:

* renal disorders
* gastrointestinal disorders
* skeletal disorders
* endocrine disorders
* drugs such as glucocorticoids , thiazide diuretics, mineral multivitamins, anti acids, tetracyclines

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10; Study Completion 2006-11

PRIMARY OUTCOMES:
serum levels of Ca, P, PTH and vitamin D metabolites and lateral chest x-ray before the treatment

SECONDARY OUTCOMES:
serum levels of Ca, P, PTH and vitamin D metabolites and lateral chest x-ray after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: parviz toossi, md, Study Chair — Skin Research Center; Hamideh Moravvej, md, Principal Investigator — Skin Research Center; Nahid Mohtasham, md, Principal Investigator — Skin Research Center
Locations (1):
- Shaheed Beheshti Medical University, Skin research center, Tehran, Iran